CLINICAL TRIAL: NCT01825707
Title: A Phase I Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-YH4808 Following Single Oral Dose Administration in Healthy Male Subjects
Brief Title: AME Study of [14C]-YH4808 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: YH4808-103
Record Dates: First submitted 2013-03-14; First posted 2013-04-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — YH4808

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C]-YH4808 200 mg (Experimental): [14C]-YH4808 200 mg
  Interventions: Drug: [14C]-YH4808 200 mg

INTERVENTIONS:
Drug: [14C]-YH4808 200 mg — [14C]-YH4808 200 mg (oral) on day1
  Other Names: YH4808 200 mg (100 µCi)

SUMMARY:
The purpose of this study is to determine the absorption, metabolism, and excretion (AME) kinetics of YH4808 and to determine and characterize metabolites present in plasma, urine, and feces in man following a single dose of [14C] YH4808 200 mg (~100 µCi ±20 µCi) administered as a single oral dose.

DETAILED DESCRIPTION:
Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to Study Entry (ie, prior to Check-in [Day -1]). Subjects will be confined at the Clinical Research Unit (CRU) from Check in (Day -1) until Discharge Criteria have been met (as early as Day 6 and as late as Day 11). In this study design, physical examinations, electrocardiograms (ECGs), vital signs, How do you feel? (HDYF?) Inquiries, and clinical laboratory evaluations will be performed at Screening, at specified times during the study, and/or at Clinic Discharge. All AEs, whether volunteered, elicited, or noted on physical examination, will be recorded throughout the study (ie, from dosing on Day 1 until Clinic Discharge [Day 11]).

ELIGIBILITY:
Inclusion Criteria:

* clinical laboratory evaluations within the reference range for the test laboratory
* negative test for selected drugs of abuse, hepatitis panel and HIV antibody screens
* able to comprehend and willing to sign an Informed Consent Form

Exclusion Criteria:

* significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs
* participation in more than 1 other radiolabeled investigational study drug trial within 12 months prior to Check-in
* donation of blood from 30 days prior to Screening through Study Completion, inclusive, or of plasma from 2 weeks prior to Screening through Study Completion, inclusive

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
PK of a single oral dose of [14C] YH4808 200 mg and its metabolites(M3, M8) | Day1-Day11
  * Maximum observed concentration in plasma, whole blood, urine, and feces
  * Time to maximum observed concentration in plasma, whole blood, urine, and feces
  * Area under the concentration-time curve from Hour 0 to the last measurable concentration
  * Assessment of Mass balance

SECONDARY OUTCOMES:
Characterization and identification of metabolites of [14C]-YH4808 in plasma, urine, and feces | Day1-Day11
assessment of the safety and tolerability of YH4808 | Day1-Day11
  * Clinical laboratory tests
  * 12-lead ECGs
  * Physical examinations
  * Vital signs
  * Adverse event assessments

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Siebers, M.D., Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States